CLINICAL TRIAL: NCT07266207
Title: A Randomized, Double-blind, Placebo-controlled Single and Multiple Ascending Dose Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetic, and Food Effects of ARD-885 Film-coated Tablets in Healthy Chinese Subjects and Patients With Rheumatoid Arthritis
Brief Title: Phase I Study to Evaluate Safety, Tolerability, Pharmacokinetic, and Food Effects of ARD-885 Film-coated Tablets in Healthy Chinese Subjects and Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Artivila (Shenzhen) Innovation Center, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KHZY-ARD885-001
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ARD-885 Tablets (Multiple Administration Dose, cohort B1~B3) (Experimental): ARD-885 Tablets, 25 mg/50 mg/100 mg, once a day(QD), from Day1~Day7
  Interventions: Drug: ARD-885 Tablets
- ARD-885 tablet (Single Administration Dose, cohort A0~A7) (Experimental): ARD-885 Tablets, 5/10/30/60/100/150/200/250 mg，a single dose on Day1
  Interventions: Drug: ARD-885 Tablets
- ARD-885 Placebo tablet (Single Ascending Dose, cohort A1~A7) (Placebo Comparator): ARD-885 Placebo tablet, a single dose on Day1
  Interventions: Drug: ARD-885 Placebo Tablet
- ARD-885 Tablets (Food Effect, cohort C1~C2) (Experimental): ARD-885 tablets, 50mg, a single dose on Day1 and Day7, fed or fasted crossover
  Interventions: Drug: ARD-885 Tablets
- ARD-885 Placebo Tablets (Multiple Administration Dose, cohort B1~B3) (Placebo Comparator): ARD-885 Placebo tablets, once a day(QD), from Day1~Day7
  Interventions: Drug: ARD-885 Placebo Tablet

INTERVENTIONS:
Drug: ARD-885 Tablets — ARD-885 Tablet is a dual-target inhibitor of IRAK4 and IRAK1.
  Arms: ARD-885 Tablets (Food Effect, cohort C1~C2); ARD-885 Tablets (Multiple Administration Dose, cohort B1~B3); ARD-885 tablet (Single Administration Dose, cohort A0~A7)
Drug: ARD-885 Placebo Tablet — Placebo Tablet to ARD-885 tablets.
  Arms: ARD-885 Placebo Tablets (Multiple Administration Dose, cohort B1~B3); ARD-885 Placebo tablet (Single Ascending Dose, cohort A1~A7)

SUMMARY:
The proposed study is a randomized, double-blind, placebo-controlled single and multiple ascending dose phase I study to evaluate the safety, tolerability, pharmacokinetic, and food effects of ARD-885 Film-coated Tablets in healthy subjects.The entire study includes 3 parts: a single ascending dose study, a multiple ascending dose study, and a food-effect bioavailability study in healthy subjects.

DETAILED DESCRIPTION:
The whole study includes 3 parts: a single ascending dose study, a multiple ascending dose study, and a food-effect bioavailability study. The SAD and MAD studies are randomized, double-blinded, and placebo-controlled studies, and the FE study is a randomized, open-label, two-period, two-treatment (2×2) crossover study.

ELIGIBILITY:
Inclusion Criteria:

* All subjects:

  1. Healthy male and female subjects of any ethnic origin between the ages of 18 and 55. Male and female patients with rheumatoid arthritis between the ages of 18 and 70.
  2. An informed consent document signed and dated by the subject. Subjects must be willing to understand and comply with all research procedures and restrictions and be able to communicate effectively with investigators.
  3. A minimum body weight of 50 kg for males and 45 kg for females, with a body mass index of 18 to 28 kg/m2 for healthy subjects and 18 to 35 kg/m2 for patients with RA.
  4. Subject (including partner) agrees to use at least one effective contraceptive method during sexual activity with partner from screening until 3 months after dosing agrees not to participate in sperm or egg donation during the study period until 3 months after the last dosing. See Section 8.1 for specific contraceptive methods.

Exclusion Criteria:

1. Known or suspected allergy to any component of ARD-885 Film-coated Tablets, or individuals with a hypersensitivity to allergies (multiple drug and food allergies), as determined by the investigator, and deemed unsuitable for inclusion.
2. Lactating women; Women of reproductive age with menstrual disorders within 90 days before administration; Women of childbearing age who have had unprotected sexual intercourse with an opposite-sex partner in the 28 days before administration. Female subjects who are lactating or have a positive serum pregnancy result during the screening period or during the trial.
3. Participated in any drug clinical trial within 90 days before administration, or the administration date of this study is still within the safety washout period specified in the previous drug clinical trial.
4. Non-physiological blood loss ≥ 200 ml within 60 days before administration (including trauma, blood collection, blood donation); Or plan to donate blood during the trial or within 30 days of administration.
5. Had a major disease that investigators considered clinically significant within 90 days before first administration; Have any active malignancy or history of malignancy in the 5 years prior to screening, with the exception of treated and considered cured skin squamous or basal cell carcinoma, cervical carcinoma in situ, or breast ductal carcinoma in situ.
6. Had major surgery within 60 days of administration, or had any surgery within 28 days of administration.
7. Infectious diseases such like fever and so on within 28 days before administration.
8. Previous use of any of the drugs or treatments listed in protocol.
9. Received vaccine or live attenuated vaccine within 1 month before administration, or who plan to receive the vaccine during the trial period.
10. Those who smoked more than 5 pieces of tobacco or equivalent daily in the 3 months before screening, or drank ≥ 14 units of alcohol per week; Or disagree with the prohibition of smoking or alcohol during the trial; Or positive alcohol serum test during screening or baseline (Day-1).
11. Those who test positive for urine drugs or have a history of drug abuse or use of drugs in the past five years.
12. +Positive for Treponema pallidum antibodies, hepatitis B surface antigen, hepatitis B core antibodies, hepatitis C virus antibodies or human immunodeficiency virus antibodies.
13. Those who is diagnosed as tuberculosis or have a history of non-tuberculous mycobacterial infections
14. Have a serious disease of the blood system or any disease that can cause hemolysis or instability of red blood cells, such as malaria, hemolytic anemia, etc..
15. At the time of screening, clinically significant gastrointestinal, liver or kidney abnormalities known abnormal which likely to affect drug intake, transport, absorption, distribution, metabolism or excretion.
16. Ingested any food or beverage containing caffein, or other xanthine-rich food or food that can induce or inhibit liver metabolic enzymes and beverages made from it within 48 hours before taking the study drug, or food or beverages containing alcohol, or other factors affecting drug absorption, distribution, metabolism, excretion, etc.
17. Those who Can not tolerate venous puncture blood collection or faint blood needle.
18. Has special requirements for diet and cannot comply with a unified diet.
19. By the investigator's decision, other factors may affect the study results and interfere with his/her participation in the study process.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AE)/Severe Adverse Events (SAE) | The first day of the first administration until 7 days after the last administration.
  Safety and tolerability are assessed by the incidence of adverse events and its severity caused by the study drug during or after dose.

SECONDARY OUTCOMES:
PK: Cmax of ARD-885. | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): Maximum observed concentration.
PK: T1/2 of ARD-885. | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): Apparent terminal elimination half-life.
PK: Tmax of ARD-885. | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): Time to reach Cmax. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value.
PK: AUC0-t of ARD-885. | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): The area under the plasma concentration-time curve from time 0 to concentration time.
PK: AUC0-last of ARD-885. | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): The area under the plasma concentration-time curve, from time 0 to the last measurable non-zero concentration.
PK: AUC0-inf of ARD-885. | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): The area under the plasma concentration-time curve from time 0 extrapolated to infinity.
PK: CL/F of ARD-885. | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): Apparent oral drug clearance.
PK: Css_max of ARD-885. | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): Steady-state maximum blood concentration in MAD study.
PK: Css_min of ARD-885. | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): Steady-state minimum blood concentration in MAD study.
PK: Tss_max of ARD-885. | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): Time to reach Cmax at steady state in MAD study.
PK: AUCss_tau of ARD-885. | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): The area under the concentration-time curve at one dosing interval after reaching a steady state in MAD study.
PK: RACmax of ARD-885. | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): Accumulation ratio on Cmax of ARD-885 in MAD study.
PK: RAAUCtau of ARD-885 | Pharmacokinetics blood samples were collected from Day1 before administration to 48 hours after the last administration.
  Pharmacokinetics (PK): Accumulation ratio on AUCtau in MAD study.
PD: The concentration of TNF-α | blood samples were collected from 1 hour before first administration to 24 hours after the last administration.
  TNF-α, IL-1β and IL-6 are a pro-inflammatory cytokines whose high expression indicating the activation of TLRs/IL-1R/NF-κB signaling pathway. Healthy Subjects in MAD study(B1~B3) will have their blood samples collected to detect levels of inflammatory factors TNF-α, IL-1β and IL-6 expression.
PD: The concentration of IL-6. | blood samples were collected from 1 hour before first administration to 24 hours after the last administration.
  TNF-α, IL-1β and IL-6 are a pro-inflammatory cytokines whose high expression indicating the activation of TLRs/IL-1R/NF-κB signaling pathway. Healthy Subjects in MAD study(B1~B3) will have their blood samples collected to detect levels of inflammatory factors TNF-α, IL-1β and IL-6 expression.
PD: The concentration of IL-1β. | blood samples were collected from 1 hour before first administration to 24 hours after the last administration.
  TNF-α, IL-1β and IL-6 are a pro-inflammatory cytokines whose high expression indicating the activation of TLRs/IL-1R/NF-κB signaling pathway. Healthy Subjects in MAD study(B1~B3) will have their blood samples collected to detect levels of inflammatory factors TNF-α, IL-1β and IL-6 expression.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Guangdong, China

IPD SHARING:
Plan to Share IPD: No